CLINICAL TRIAL: NCT06276387
Title: Defining Stress REsilience And Mindfulness Effects in Rheumatoid Arthritis
Acronym: DREAMER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: K23AT011768-01 (NIH); K23AT011768 (NIH)
Record Dates: First submitted 2024-02-16; First posted 2024-02-26 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Arthritis, Rheumatoid
Keywords: Mindfulness; Rheumatic Diseases; Autoimmune Diseases
MeSH Terms: conditions — Arthritis, Rheumatoid; Rheumatic Diseases; Autoimmune Diseases | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to participate in a mindfulness-based stress reduction (MBSR) course or treatment as usual (TAU). Randomization will be done using a program-tracking system.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Physicians completing joint exams to assess clinical disease activity, including the principal investigator, will be blinded to participant assignment. It will not be possible for participants to be blinded to treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Program (Experimental): Individuals in the mindfulness group will complete an 8-week mindfulness course that has been adapted for individuals with rheumatic diseases (MBSR-RD).
  Interventions: Behavioral: Mindfulness Program
- Treatment as Usual (TAU) (No Intervention): Individuals in the TAU group will continue engaging in routine care and be asked to refrain from participating in mindfulness programs during the trial.

INTERVENTIONS:
Behavioral: Mindfulness Program — Participants will receive eight weekly 2.5-hour group sessions and one day-long silent retreat, delivered online. Intervention content will include the MBSR program, which has been extensively studied with many different chronic conditions, and augmentations for individuals with rheumatic diseases. Each MBSR session will include meditation practices (e.g., sitting meditation, body scan, gentle hatha yoga, walking meditation, mindfulness of daily activities, awareness of pleasant and unpleasant events) and review of home practice. Participants will complete daily home practices for about 45 minutes per day and log their practice.
  Other Names: Mindfulness-Based Stress Reduction; MBSR; MBSR-RD
  Arms: Mindfulness Program

SUMMARY:
This clinical trial will test a mindfulness program in individuals with rheumatoid arthritis (RA). The main goals of this pilot study are to:

* Assess patient satisfaction with a mindfulness course
* Identify barriers to participation in, or completion of, a mindfulness course
* Gather initial information to understand how a mindfulness course impacts RA symptoms

Participants will:

* Complete online questionnaires
* Attend two in-person study visits, involving a brief joint exam and blood draw
* Roughly half the participants will have the chance to participate in an 8-week online mindfulness course
* Roughly half the participants will be invited to participate in an online focus group following completion of the mindfulness course

Researchers will compare those in the mindfulness course with those receiving standard care in preparation for a larger future study to see how mindfulness impacts stress and inflammation in individuals with RA.

DETAILED DESCRIPTION:
Participants will complete an initial eligibility screening, and if they are eligible, they will meet with a study staff member to review study procedures and answer any questions they might have about participating. If they would like to participate following this meeting, they will provide written consent and be enrolled in the study. Following enrollment, participants will complete an in-person study visit that will last up to one hour and include a brief joint exam, blood draw, and questionnaires. After this study visit, they will be randomly assigned to "treatment-as-usual" (TAU) or the mindfulness group. If assigned to the mindfulness group, they will participate in an 8-week online mindfulness course and online focus group following the course. All participants will complete a final in-person study visit at the end of the study, which will mimic the procedures of the first study visit.

ELIGIBILITY:
Inclusion Criteria:

* Physician-confirmed diagnosis of rheumatoid arthritis (RA)
* Access to a web-enabled computer, smartphone, or tablet

Exclusion Criteria:

* RA disease activity in remission
* Current regular mindfulness practice (> 20 minutes per week)
* Inability to participate in an intensive 8-week online mindfulness course
* Prior participation in a mindfulness-based stress reduction (MBSR) course

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-22 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction as Assessed by CSQ-8, Adapted for DREAMER Study | 8 weeks
  A modified version of the 8-item Client Satisfaction Questionnaire (CSQ-8) will be used to evaluate acceptability of the mindfulness program by patients in the treatment group. A few of the words in the original CSQ-8 were changed to make the questions relevant to the mindfulness program. Scores on the CSQ-8 range from 8-32, with higher scores indicating greater satisfaction. Scores ≥ 24 indicate adequate satisfaction.

SECONDARY OUTCOMES:
MBSR Course Attendance (Intervention Adherence) | 8 weeks
  Intervention adherence will be operationalized as the percentage of participants who were randomized to the mindfulness group and attended at least six of the eight group sessions.
Percent of Study Completers (Study Retention) | 8 weeks
  Study retention will be operationalized as the number of participants who completed assessments (questionnaires and physician disease activity assessment) at the follow-up time-point divided by the number of participants who enrolled in the study, multiplied by 100.

OTHER OUTCOMES:
Clinical Disease Activity Index (CDAI) | 8 weeks
  The CDAI, is a patient and provider composite tool that incorporates data from the patient global assessment, provider global assessment, 28 swollen joint count, and 28 tender joint count. It is a validated measure of RA disease activity that is recommended by the American College of Rheumatology for use in clinical practice and RA pharmaceutical trials. This is an exploratory outcome measure as the current study is not adequately powered to assess whether MBSR-RD is effective for improving clinical outcomes.
Disease Activity Score in 28 Joints (DAS-28) | change from baseline to 8 weeks
  The DAS-28 is a validated measure of disease activity that is frequently employed in RA pharmaceutical clinical trials. It incorporates data from the patient global assessment, provider global assessment, 28 swollen joint count, 28 tender joint count, and a laboratory measure of systemic inflammation from either the erythrocyte sedimentation rate (ESR) or c-reactive protein (CRP). This is an exploratory outcome measure as the current study is not adequately powered to assess whether MBSR-RD is effective for improving clinical outcomes.
Modified Rheumatoid Arthritis Disease Activity Index, 5-item (RADAI-5) | change from baseline to 8 weeks
  The RADAI-5 is a validated patient-reported assessment of RA disease activity that comprises five questions in a Likert format from 0 to 10. We will use a modified version of the RADAI-5 in which the period of recall is 2 weeks instead of 6 months. This is an exploratory outcome measure as the current study is not adequately powered to assess whether MBSR-RD is effective for improving clinical outcomes.
Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference, 4-Item Scale | change from baseline to 8 weeks
  The PROMIS Pain Interference scale measures the extent to which pain hinders an individual's engagement with physical, mental, cognitive, emotional, recreational, and social activities. This is an exploratory outcome measure as the current study is not adequately powered to assess whether MBSR-RD is effective for improving clinical outcomes.
Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue, 4-Item Scale | change from baseline to 8 weeks
  The PROMIS Fatigue scale measures the experience of fatigue and associated impact on daily life. This is an exploratory outcome measure as the current study is not adequately powered to assess whether MBSR-RD is effective for improving clinical outcomes.
Patient-Reported Outcomes Measurement Information System (PROMIS) Global Mindfulness, 13-item Scale | change from baseline to 8 weeks
  The PROMIS Mindfulness scale measures the capacity for present moment awareness. This is an exploratory outcome measure and will be used to determine whether mindfulness mediates improvements in clinical outcomes such as pain among participant in the active treatment group.
Perceived Stress Scale, 10-item | change from baseline to 8 weeks
  The perceived stress scale measures general perceptions of the degree to which situations in one's life are viewed as stressful. This is an exploratory outcome measure and will be used to determine whether changes in perceived stress mediate improvements in clinical outcomes such as pain among participant in the active treatment group.
Brief Resilience Scale | change from baseline to 8 weeks
  The Brief Resilience Scale measures the perceived ability to bounce back or recover from stress. This is an exploratory outcome measure and will be used to determine whether stress resilience mediates improvements in clinical outcomes such as pain among participant in the active treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L Patterson, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Osher Center for Integrative Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No